CLINICAL TRIAL: NCT07268768
Title: Personological Structure, Cognitive Functions and Central Sensitization in Headache: Obstacles and Resources in the Treatment of Chronic and Episodic Headache.
Brief Title: PERSONOLOGICAL STRUCTURE, COGNITIVE FUNCTIONS AND CENTRAL SENSITIZATION IN HEADACHE
Acronym: AURA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Anna Anselmo, Psychologist, IRCCS Centro Neurolesi Bonino Pulejo
Other Study IDs: CEL/U117/25
Record Dates: First submitted 2025-11-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic and Episodic Headache; Headache Disorders
Keywords: chronic migraine; central sensitization; cognitive impairment; personality disorders; treatment adherence; anxiety; depression;
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Headache Disorders; Cognitive Dysfunction; Personality Disorders; Treatment Adherence and Compliance; Anxiety Disorders; Depression | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic headache: Patients suffering from chronic headache
  Interventions: Other: Neuropsychological assessment
- Episodic headache: Patients suffering from episodic headache
  Interventions: Other: Neuropsychological assessment

INTERVENTIONS:
Other: Neuropsychological assessment — Standardized and ad hoc test battery for comprehensive neuropsychological assessment

SUMMARY:
Headache, in its episodic and chronic forms, cannot be considered solely as an isolated neurological symptom, but as a complex condition of a bio-psycho-social nature. While in the episodic form the painful episodes occur intermittently and have a variable impact on daily life, in the chronic form the disease evolves towards persistent pain, with more significant consequences on personal, social and work functioning. The following study protocol aims to investigate in an integrated manner the neurological, cognitive and psychological mechanisms involved in headache, with particular attention to the differences between episodic and chronic forms. The main objective is to assess the neuropsychological profiles and pain response of patients, monitoring their evolution over a period of approximately six months, considering the impact of central sensitisation, personality structure and any psychopathological comorbidities on pain management and treatment adherence. The protocol adopts a multidimensional approach aimed at optimising therapeutic efficacy and improving patients' quality of life, preventing progression to chronicity.

DETAILED DESCRIPTION:
This is an observational, prospective study with two assessment timepoints: baseline (T0) and follow-up at approximately six months (T1). The overall duration of the project is estimated at about three years, including enrollment of all planned participants, completion of follow-up, data analysis and dissemination of results.

The study is conducted at the IRCCS Centro Neurolesi "Bonino-Pulejo" with UTIC P.O. "Piemonte" in Messina, Italy, within the Headache Outpatient Clinic.

The target population consists of adult patients with a diagnosis of chronic or episodic headache referring to the Headache Outpatient Clinic. Sample size was calculated using G*Power 3.1, taking as reference the primary objective of comparing the evolution (baseline vs T1) of main clinical-neuropsychological outcomes between chronic and episodic headache groups. The primary test was modeled as a repeated-measures ANOVA on the group×time interaction (two groups, two measurements), analogous to the interaction component of a linear mixed model.

With a significance level α = 0.05, statistical power 1-β = 0.90, intra-subject correlation r = 0.60 and two measurements, assuming an interaction effect size f = 0.20 and nonsphericity correction ε = 1, the minimum required sample size is N = 56 subjects (28 per group). Taking into account an expected dropout rate of 15%, the required enrollment was increased to N = 64 participants (32 per group), in order to preserve the planned power for the primary analysis.

Inclusion criteria

* Age between 18 and 60 years;
* Diagnosis of chronic or episodic headache;
* Patients attending the Headache Outpatient Clinic. Exclusion criteria
* Presence of severe psychiatric and neurological disorders;
* Presence of oncological diseases in terminal stage Identification and numbering of subjects In accordance with Good Clinical Practice (GCP), each subject is identified by an unequivocal numerical code that serves as the subject's identifier throughout the study. In this protocol, the code consists of a three-digit subject number assigned in progressive order starting from 001 when the subject signs the informed consent form. The investigator records the subject's name and corresponding code in a dedicated dataset accessible only to authorized study collaborators, thereby ensuring traceability and confidentiality.

Study procedures All potentially eligible subjects are informed about the aims and procedures of the study and are free to choose whether to participate. Only after the subject, or his/her legal representative, has agreed to participate and has signed the informed consent form, do the investigators proceed with the planned activities.

Clinical data for each subject are stored in a secure database accessible to study collaborators via personal credentials. After verifying the inclusion and exclusion criteria and obtaining informed consent, patients are formally enrolled and scheduled for the baseline assessment (T0).

Baseline visit (T0)

At T0, the following procedures are performed:

* Verification of inclusion and exclusion criteria
* Collection of demographic data
* Collection of clinical history, including headache characteristics, comorbidities and medication use

After the clinical assessment, a standardized battery of tests is administered to evaluate dimensions related to chronic pain and quality of life:

* Cognitive functions: Brief Cognitive Status Exam (BCSE) and/or Montreal Cognitive Assessment (MoCA)
* Pain intensity and central sensitization: Numeric Pain Rating Scale (NPRS) and Central Sensitization Inventory (CSI)
* Personality: Minnesota Multiphasic Personality Inventory 3 (MMPI-3)
* Treatment engagement and adherence: Patient Health Engagement Scale (PHE-S) and Morisky Medication Adherence Scale (MMAS)
* Psychological distress: Beck Depression Inventory (BDI) and State-Trait Anxiety Inventory (STAI)
* Digital habits: ad-hoc questionnaire on digital behaviors in patients with headache

Follow-up visit (T1) At approximately six months (T1), patients return for follow-up. All standardized instruments administered at T0 are readministered in order to evaluate changes over time in cognitive functioning, pain intensity and sensitization, personality and psychopathological dimensions, treatment adherence and digital habits.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years;
* Diagnosis of chronic or episodic headache;
* Patients attending the Headache Outpatient Clinic.

Exclusion Criteria:

* Presence of severe psychiatric and neurological disorders;
* Presence of oncological diseases in terminal stage

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The target population consists of adult patients with a diagnosis of chronic or episodic headache referring to the Headache Outpatient Clinic. Sample size was calculated using G*Power 3.1, taking as reference the primary objective of comparing the evolution (baseline vs T1) of main clinical-neuropsychological outcomes between chronic and episodic headache groups. The primary test was modeled as a repeated-measures ANOVA on the group×time interaction (two groups, two measurements), analogous to the interaction component of a linear mixed model.
  With a significance level α = 0.05, statistical power 1-β = 0.90, intra-subject correlation r = 0.60 and two measurements, assuming an interaction effect size f = 0.20 and nonsphericity correction ε = 1, the minimum required sample size is N = 56 subjects (28 per group). Taking into account an expected dropout rate of 15%, the required enrollment was increased to N = 64 participants (32 per group), in order to preserve the planned power for the p
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-11-20 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological assessment | 6 months
  •Cognitive functions: Brief Cognitive Status Exam (BCSE) and/or Montreal Cognitive Assessment (MoCA)

SECONDARY OUTCOMES:
Central sensitization | 6 months
  Central Sensitization Inventory (CSI)

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Centro Neurolesi Bonino Pulejo, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No